CLINICAL TRIAL: NCT00302861
Title: Phase 1/2 Study to Evaluate the Feasibility and Tolerability of Treatment of Previously Untreated B-CLL Chronic Lymphocytic Leukemia (B-CLL) Patients With Recombinant Idiotype Conjugated to KLH (Id-KLH) Administered With GM-CSF
Brief Title: A Study to Evaluate the Treatment of Previously Untreated B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genitope Corporation (Industry)
Other Study IDs: 2005-11; NCT00313651 (obsolete NCT alias)
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: B-Cll
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Biological: MyVax

SUMMARY:
This is a multi-center, open-label, single arm Phase 1/2 study evaluating the feasibility, safety, and tolerability of a series of 16 immunizations of Id-KLH with GM-CSF in patients with previously untreated B-CLL. The length of the controlled portion of the study is two years. The study will be conducted at investigative sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Have signed a written informed consent
* B-CLL diagnosis
* Rai Stage 0, I, or II
* Previously untreated
* Be able to watch and wait for approximately 8 months following submission of blood (or tissue) while Id-KLH is being manufactured

Exclusion Criteria:

* Anti-leukemia treatment prior to beginning immunization
* Anti-leukemia treatment other than Id-KLH during immunizations
* Prior malignancy (excluding basal cell carcinoma and cervical carcinoma in situ)
* Pregnant or lactating
* Patients with known autoimmune disease (including previously treated autoimmune hemolytic anemia or immune thrombocytopenia)
* Participation in any other clinical trial in which an investigational agent is administered

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2006-03

PRIMARY OUTCOMES:
The proportion of patients with positive humoral immune responses
Safety and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kipps, M.D., Principal Investigator — University of California, San Diego